CLINICAL TRIAL: NCT03358108
Title: A Prospective, Multicentre Observational Follow-up Study of PegIFN Treatment Sustained Response in Nucleoside Experienced Patients With Chronic Hepatitis B (the OCEAN Study)
Brief Title: A Prospective,Observational Follow-up Study of Nucleoside Treated Patients With Chronic Hepatitis B (OCEAN Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: OCEAN study
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: interferon group: formerly interferon group (including interferon alone or interferon combined with other drugs)
- Group B:nucleoside analogue group: formerly nucleoside analogue treatment group. Each group was followed for five years

SUMMARY:
This is a prospective, multicentre observational follow-up study of PegIFN treatment unstained response in nucleoside experienced patients with Chronic Hepatitis B.Patients will join this study after finished following clinical trail about A Study of Combination or Sequential Treatment With PEGASYS (Peginterferon Alfa-2a) and Entecavir in Patients With HBeAg Positive Chronic Hepatitis B(OSST trail),A Real-World Study of Pegylated Interferon In Nucleoside-treated Patients With Chronic Hepatitis B (COST study), Combination Therapy With Interferon Plus Interleukin 2 and Hepatitis B Vaccine in Chronic Hepatitis B Patients(Endeavor study),A Prospective Clinical Trial in Chronic Hepatitis B Patients Nucleotide Analogues Experienced (Anchor A Study),Sequential/Combination Therapy in Nucleoside or Nucleotide Analogue (NA)-Suppressed Chronic Hepatitis B Patients (NPGV study).We plan to compare the HBsAg negative rate and maintenance rate,the occurrence of liver cirrhosis and the occurrence rate of hepatocellular carcinoma(HCC) related to hepatitis B virus(HBV) within five years between interferon group (including interferon alone or interferon combined with other drugs) and nucleoside analogues.Patients were divided into two groups based on whether they received interferon or not.

DETAILED DESCRIPTION:
Patients who treated with nucleoside analogs, and previously took part in the OSST,COST,Endeavor, Anchor NPGV studies, were included in the observational study after they finished. The patients entered the following two observation groups based on previous studies: Group A: formerly interferon group (including interferon alone or interferon combined with other drugs); Group B: formerly nucleoside analogue treatment group. Each group was followed for five years.All patients were followed up for physical examination (vital signs, whole body examination) and laboratory assessment (HBsAg quantification, HBeAg quantification, HBV DNA, HBV immunology marker, blood routine, blood biochemistry, alpha fetoprotein, Fibroscan, liver Doppler) in every six month.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. Have finished the OSST,COST,Endeavor, Anchor,NPGV studies;
3. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. patients have not participated in the OSST,Cost,Endeavor,Anchor or NPGV study ;
2. unable or unwilling to provide informed consent or follow the research requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who treated with nucleoside analogs, and previously took part in the OSST,COST,Endeavor, Anchor,NPGV studies, were included in the observational study after they finished.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg negative at week 260 | week 260
  Compare the HBsAg negative rate at week 260 with that at baseline

SECONDARY OUTCOMES:
The maintenance response rate of HBsAg negativity at week 260 | week 260
  the proportion of patients with sustained HBsAg negativity at week 260 among the patients whose HBsAg negative at baseline
HBsAg quantification decline from baseline to week 260 | week 260
  HBsAg quantification decline from baseline to week 260 are measured.
Change from baseline in HBsAg seroconversion at week 260 | week 260
  HBsAg seroconversion from baseline is measured
The rate of HBsAb positive at week 260 | week 260
  Compare the rate of HBsAb positive at week 260 with that at baseline
Measure the Fibroscan value | week 260
  Fibroscan value from baseline is measured
the occurrence rate of liver cirrhosis | week 260
  Statistics for occurrence rates of liver cirrhosis
the occurrence rate of HCC related to HBV | week 260
  Statistics for occurrence rates of HCC related to HBV
The proportion of patients with HBV DNA <1000 copies / mL | week 260
  Statistics the proportion of patients with HBV DNA <1000 copies / mL

CONTACTS AND LOCATIONS:
Overall Officials: Ning Qin, Doctor, Principal Investigator — Department of Infectious Diseases, Tongji Hospital
Locations (11):
- China (11):
  - BeiJing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Zhejiang, Hangzhou
  - Tongji Hospital, Wuhan, Hubei
  - Departmen of infectious disease, Xiangya Hospital, Central-south Universit, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Traditional Chinese Medicine,Xiamen Hospital, Shantou, Xiamen
  - The first affiliated hospital of Wenzhou medical universtiy, Wenzhou, Zhejiang